CLINICAL TRIAL: NCT03716323
Title: Evaluation of Marginal Bone Loss After Immediate Implant Placement in Maxillary Premolar Zone With Allograft Versus Xenograft
Brief Title: Immediate Implants in Maxillary Premolar Region Using Xenograft vs Allograft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Abdallah AbdelFattah, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CairoMOImplant
Record Dates: First submitted 2018-10-21; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Badly Broken Maxillary Premolars Indicated for Extraction
MeSH Terms: interventions — Transplantation, Heterologous; Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- immediate premolar implant with xenograft and allograft (Experimental): Immediate Implant Placement in Maxillary Premolar zone with grafting the jumping gap using xenograft and allograft
  Interventions: Device: immediate premolar implant with xenograft and allograft

INTERVENTIONS:
Device: immediate premolar implant with xenograft and allograft — * A peritome will be used for atraumatic extraction of remaining roots.
  * The extraction socket will be evaluated for absence of any fenestration or granulation tissues.
  * Copious normal saline irrigation and curettage will be performed.
  * In the study group: Immediate implant insertion following standard manufacturer's recommended surgical protocol followed by grafting the jumping gap with cortico-cancellous allograft (MinerOss®, BioHorizons, USA)
  * In the control group: Immediate implant insertion following standard manufacturer's recommended surgical protocol followed by grafting the jumping gap with anorganic bovine bone mineral xenograft (Bio-Oss®, Geistlich, USA)

SUMMARY:
Immediate implant placement has the disadvantage of difficulty in obtaining primary stability, lack of adequate soft tissue coverage and also the control of the implant position is difficult in addition to the cost of the graft. Autogenous bone graft is considered to be the golden standard for grafting as it has osteoconductive , osteoinductive and osteogenic functions , however it has the problems of donor site morbidity , the need for two surgeries as well as post operative swelling and discomfort of the patient , so alternative bone grafts as allografts and xenografts, has been introduced.

DETAILED DESCRIPTION:
Allograft bone is obtained from individuals of the same species, derived from human-cadaver bone that has been selected and tested to be free of HIV and transmitted diseases. The most common allograft used is dematerialized freeze-dried bone allograft (DFDBA), provide type I collagen, which comprises most of the organic component of bone. In addition, allograft contains BMPs, which stimulate osteoinduction. There are thirteen proteins have been identified (BMP1-BMP13) which are osteoinductive compounds and stimulate new bone formation. A previous study demonstrated that, a combination of osseous coagulum collected during preparation and freeze-dried bone allograft placed at immediate implant insertion and loading. Xenografts are one of the most successful and widely used grafting materials nowadays as a replacement for autogenous bone grafts. Studies showed that xenografts are very successful because of their osteoconductive properties, their denisty which provides stabilization to the graft and implant and they supply the necessary minerals for bone formation as xenograft don't resorb completely.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with badly broken teeth in upper premolar zone indicated for extraction, presence of at least 3 mm of bone beyond the root apex to guarantee implant primary stability, implant placement within the alveoli confines.
* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* Presence of fenestrations or dehiscence of the residual bony walls after extraction.
* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Marginal Bone Loss | 6 months
  The amount of marginal bone loss will be measured using cone beam computed tomography